CLINICAL TRIAL: NCT04528134
Title: The Effect of Light-cured Fluoride Varnish to Remineralize Post-orthodontic White Spot Lesions and Change the Oral Microbiome: a Double-blind, Split-mouth Randomized Clinical Trial
Brief Title: Orthodontic Varnish Microbiology Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Tyler Brennan, Orthodontic Resident, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB#20-001077
Record Dates: First submitted 2020-06-12; First posted 2020-08-27 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Dental Caries; Dental Plaque; Dental White Spot
Keywords: Orthodontics
MeSH Terms: conditions — Dental Caries; Dental Plaque

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized into one of 3 groups, each of which will receive two of the following three interventions: extended contact varnish, traditional fluoride varnish, placebo varnish. Subjects will receive the interventions in a split-mouth design, with one treatment on half of their teeth and another treatment on the other half of their teeth.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not know which interventions they receive. The investigator, who will be providing the treatment, will be aware of which treatments they are receiving (the investigator is impossible to mask due to the different applications of the treatment interventions). Outcomes assessors will be masked and score outcomes based on photos and microbiological data that is de-identified.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Extended Contact RMGI Varnish/5% Sodium Fluoride Varnish (Experimental): This group will receive extended contact (XT) varnish on their upper left and lower right teeth, and traditional 5% sodium fluoride varnish on their upper right and lower left teeth.
  Interventions: Device: Extended Contact RMGI (Resin-modified Glass Ionomer) Varnish; Device: 5% Sodium Fluoride Varnish
- Placebo Varnish/Extended Contact RMGI Varnish (Experimental): This group will receive placebo varnish on their upper left and lower right teeth, and extended contact (XT) varnish on their upper right and lower left teeth.
  Interventions: Device: Extended Contact RMGI (Resin-modified Glass Ionomer) Varnish
- 5% Sodium Fluoride Varnish/Placebo Varnish (Active Comparator): This group will receive traditional 5% sodium fluoride varnish on their upper left and lower right teeth, and placebo varnish on their upper right and lower left teeth.
  Interventions: Device: 5% Sodium Fluoride Varnish

INTERVENTIONS:
Device: Extended Contact RMGI (Resin-modified Glass Ionomer) Varnish — This is a light-cured, durable coating that forms an immediate layer of protection that releases fluoride, calcium and phosphate and can be recharged with fluoride by using fluoride-containing products over the 6-month life of the product.
  Other Names: 3M™ Vanish™ XT Extended Contact Varnish
  Arms: Extended Contact RMGI Varnish/5% Sodium Fluoride Varnish; Placebo Varnish/Extended Contact RMGI Varnish
Device: 5% Sodium Fluoride Varnish — This is a 5% Sodium Fluoride varnish that hardens on the teeth upon contact with saliva.
  Other Names: Henry Schein Acclean 5% Sodium Fluoride Varnish
  Arms: 5% Sodium Fluoride Varnish/Placebo Varnish; Extended Contact RMGI Varnish/5% Sodium Fluoride Varnish

SUMMARY:
Orthodontic treatment is common in teenagers, which typically involve the attachment of metal brackets to the teeth. These brackets often impede proper oral hygiene, leading to plaque accumulation and the development of white spots lesions (the early stage of cavity development). Our study aims to investigate the efficacy of different commercially available fluoride varnishes to treat these white spot lesions after the completion of orthodontic treatment and evaluate their effect on the oral microbiome.

Target enrollment is 120 subjects. The study will follow a split-mouth design, with each subject receiving different treatment on the left and right sides of their mouth. The subjects will be randomized into 3 groups, with each group receiving two of the following three options: placebo varnish, traditional sodium fluoride varnish, and a resin-modified glass ionomer light-cured fluoride varnish. There will be 4 total visits for this study:

Baseline (day 0): Oral health assessed, plaque collected, intraoral photos taken, dental cleaning performed, DiagnoDent measurements taken, varnishes applied T1 (day 30): Oral health assessed, plaque collected, intraoral photos taken, DiagnoDent measurements taken, varnishes reapplied T2 (day 90): Oral health assessed, plaque collected, intraoral photos taken, DiagnoDent measurements taken, varnishes reapplied T3 (day 180): Oral health assessed, plaque collected, intraoral photos taken, DiagnoDent measurements taken, dental cleaning performed

Participants will be instructed to use regular fluoridated toothpaste and floss twice per day for the duration of the study.

DETAILED DESCRIPTION:
1. Orthodontic patients ages 12-27 (target 120 subjects) nearing the end of treatment with metal braces at the UCLA Orthodontic Clinic will be recruited.
2. Patients will be consented by the investigators or an eligible and trained orthodontic resident.
3. Participants will be assigned into one of three groups via stratified permuted block randomization. The groups will receive treatment as follows in a split-mouth study design:

   Group 1 - extended contact varnish on upper left and lower right teeth, 5% fluoride varnish on upper right and lower left teeth Group 2 - placebo varnish on upper left and lower right teeth, extended contact varnish on upper right and lower left teeth Group 3 - 5% fluoride varnish on upper left and lower right teeth, placebo varnish on upper right and lower left teeth
4. Shortly after a subject's braces are removed, each subject will fill out an oral health questionnaire and the investigators will use Trace Plaque Disclosing Liquid (a safe, commercially available product) to visualize the plaque. Intraoral photos of only the teeth surfaces will be taken. Dental plaque samples will be collected from buccal surfaces of the teeth. The plaque will be collected with a sterile dental instrument and carefully deposited into a sterile plastic collection tube containing a nutrient solution for the bacteria. After collection, the samples will be taken to the laboratory for further analysis and no subject identifiers will be used. The samples will be plated and total DNA from each will be extracted, and sequencing analysis will be performed in order to determine the relative abundance of each species in the samples.
5. A professional cleaning will be done of the subjects teeth to remove all remaining plaque and calculus buildup on the teeth.
6. After the cleaning, the subject will rinse with water and a second set of intraoral photos will be taken. The teeth will then be air dried for 15 seconds, and a third set of intraoral photos will be taken.
7. The extent of the demineralized white spot lesions will be quantitatively assessed using the DiagnoDent, where a laser is shined on the teeth and the fluorescence is measured to assess the depth/severity of the demineralization.
8. The study varnishes will be applied to the patient's teeth (according to the manufacturer's instructions), consistent with their group allocation.
9. The patient will be given written post-op instructions, including oral hygiene instructions to use OTC sodium fluoride toothpaste and a manual toothbrush. The subjects will be asked to refrain from using adjunctive fluoride products (such as mouthwash) for the duration of the study. Since all subjects will receive another professional cleaning at their 6-month visit (consistent with the standard of care to receive professional cleanings every 6 months), they will be asked to not receive additional dental cleanings from outside providers.
10. Subjects will return to the clinic after 30, 90, and 180 days. At each appointment, they will have their plaque disclosed with Trace Plaque Disclosing solution, have 3 sets of intraoral photos taken (with plaque, with clean/moist teeth, and with clean/dry teeth), have the white spot lesion severity measured with the DiagnoDent, and have the varnishes reapplied to their teeth (except at the last, where the varnish will not be reapplied).
11. At the final visit (day 180), subjects will receive a professional dental cleaning after the photos have been assessed.
12. After study completion, blinded investigators will use the intraoral photos to (1) assess the extent of plaque using various plaque indices, and (2) assess the severity of white spot lesions using various visual indices.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 12-17 years of age, inclusive, at the time the Assent and Informed Consent Form is signed
* Systemically healthy, as determined by the investigator (in consultation with the Medical Monitor, as needed), based on medical history, concurrent illnesses, laboratory results, concomitant medications, oral cavity assessment, and targeted physical examination (extraoral, head and neck) during screening
* Is approaching the end of their orthodontic treatment using metal fixed oral appliances (brackets) on at least the maxillary arch
* Subject has at least two visible white spot lesions at the time of recruitment on teeth treated with fixed oral appliances
* Subject is willing to use only oral care products that fall within the standard of care (manual toothbrush and sodium fluoride toothpaste) for the duration of the study.
* Subject is willing to postpone dental cleanings between the baseline and final visit (since subjects will receive cleanings 6 months apart at both the baseline and final visit, the standard of care will be maintained).
* Subject is willing and able to comply with oral hygiene and diet instructions.
* Subject is able to understand and sign the Assent and/or Informed Consent Form prior to initiation of study procedures
* Subject is able to communicate with the Investigator/study personnel, understand and comply with the study requirements, and is willing to return for protocol-specified visits at the appointed times.

Exclusion Criteria:

* Advanced periodontal disease
* Medical condition (e.g. artificial heart valve, history of infective endocarditis, cardiac transplant with valvular dysfunction, congenital heart disease or total joint replacement) for which antibiotics are recommended prior to dental visits and/or procedures
* Pathologic lesions of the oral cavity (suspected or confirmed)
* Use of systemic antibiotics, topical oral antibiotics, or use of other drugs, which in the opinion of the investigators could influence the study outcome, within 30 days prior to screening.
* Presence of any condition or concurrent illness, which in the opinion of the investigators, would compromise normal immune function ((e.g., diabetes, rheumatoid arthritis, lupus, liver disease, organ transplant, etc.), interfere with the use of study dentifrice and oral care products, or interfere with the ability to comply with study requirements, or jeopardize the safety of the subject or the validity of the study results
* Presence of xerostomia (dry mouth).

Ages: 12 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
White Spot Lesion severity | 6 months
  Assessed change in severity of white spots on the teeth as measured by the DiagnoDent, which uses quantitative light-induced fluorescence to assess the depth/severity of enamel demineralization.

SECONDARY OUTCOMES:
Dental Plaque Levels | 6 months
  Assessed change in plaque levels, as measured by the Turesky-modified Quigley Hein Plaque Index.
Microbiome Composition | 6 months
  Change in microbial composition of dental plaque, as measured by sequencing of the 16s rRNA gene.
Plaque and Saliva Microbial Colonization | 6 months
  Change in amounts of Streptococcus mutans and Candida albicans, as measured by counting Colony-Forming Units (CFUs) after plating saliva samples.
White Spot Lesion Clinical Appearance | 6 months
  Assessed change in the visual appearance of white spots on the teeth, as measured by a Visual Index from clinical photographs.
Salivary flow rate | 6 months
  Assessing saliva flow at rest and when stimulated by chewing by time it takes for salivary droplets to form on the lower lip and how long it takes to expectorate 5mL of saliva.
Salivary pH | 6 months
  Assessing resting and stimulated saliva pH by using pH strips dipped in saliva samples.
Saliva Buffering Capacity | 6 months
  Assessing saliva buffering capacity using a test strip onto which drops of stimulated saliva is dropped with a pipette.
Saliva Consistency | 6 months
  Semi-qualitative assessment of saliva consistency while resting in the mouth - Normal viscosity (Watery/clear), Increased viscosity (Frothy/bubbly), High viscosity (Sticky/frothy)

CONTACTS AND LOCATIONS:
Overall Officials: Tyler Brennan, DDS, Principal Investigator — University of California, Los Angeles; Renate Lux, PhD, Study Chair — University of California, Los Angeles; Nini Tran, DDS, PhD, Study Director — University of California, Los Angeles
Locations (1):
- UCLA School of Dentistry, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
Only de-identified and aggregate data will be made available to researchers outside the study team.

REFERENCES:
- [Background] Klaus K, Eichenauer J, Sprenger R, Ruf S. Oral microbiota carriage in patients with multibracket appliance in relation to the quality of oral hygiene. Head Face Med. 2016 Oct 28;12(1):28. doi: 10.1186/s13005-016-0125-x. PMID 27793169
- [Background] Freitas AO, Marquezan M, Nojima Mda C, Alviano DS, Maia LC. The influence of orthodontic fixed appliances on the oral microbiota: a systematic review. Dental Press J Orthod. 2014 Mar-Apr;19(2):46-55. doi: 10.1590/2176-9451.19.2.046-055.oar. PMID 24945514
- [Background] Sundararaj D, Venkatachalapathy S, Tandon A, Pereira A. Critical evaluation of incidence and prevalence of white spot lesions during fixed orthodontic appliance treatment: A meta-analysis. J Int Soc Prev Community Dent. 2015 Nov-Dec;5(6):433-9. doi: 10.4103/2231-0762.167719. PMID 26759794
- [Background] Tasios T, Papageorgiou SN, Papadopoulos MA, Tsapas A, Haidich AB. Prevention of orthodontic enamel demineralization: A systematic review with meta-analyses. Orthod Craniofac Res. 2019 Nov;22(4):225-235. doi: 10.1111/ocr.12322. Epub 2019 May 27. PMID 31081584
- [Background] Mehta A, Paramshivam G, Chugh VK, Singh S, Halkai S, Kumar S. Effect of light-curable fluoride varnish on enamel demineralization adjacent to orthodontic brackets: an in-vivo study. Am J Orthod Dentofacial Orthop. 2015 Nov;148(5):814-20. doi: 10.1016/j.ajodo.2015.05.022. PMID 26522042